CLINICAL TRIAL: NCT02880969
Title: Effect of Individual and Populational Determinants on End Stage Renal Disease Children Quality of Life, During Dialysis Period.
Acronym: CQFD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-22; 2012-A00761-42 (Other: Ansm)
Record Dates: First submitted 2016-08-12; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Kidney Dysfunctions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with end stage renal disease undergoing dialysis (Experimental)
  Interventions: Behavioral: answering questionnaires

INTERVENTIONS:
Behavioral: answering questionnaires

SUMMARY:
End stage renal disease (ESRD) is a severe pathology, treated by dialysis on standby of graft availability. Being under dialysis requires a recourse to pluri-weekly magazine of health care system, impacting negatively patient's quality of life (QoL) and their entourage, at a psychological, physical and social level.

Although further studies have assessed QoL in ESRD grafted children, a lack of information exists concerning patients' QoL during dialysis before graft. In addition, some limits could be listed, these studies have small samples, 50 patients at all, and only clinical determinants are studied. A larger clinical research assessing children's QoL studying individual and populational factors is necessary.

The aim of the study is to assess the influence of individual and populational determinants on children's QoL with ESRD, treated by dialysis.

Material & Method An exhaustive inclusion of patient with ESRD treated by dialysis will be realized at 20 French Pediatrics Dialysis Centers. Inclusion criteria are i) two genders, ii) younger than 18 years old, iii) having an ESRD treated by dialysis, iv) attending at one of the French Pediatrics Dialysis Centers for treatment between the 1st September 2012 and the 31th August 2014, v) being at their fourth to sixth week of dialysis. Patients will be re-evaluated at 4th month and 7th month after first dialysis. Informed consent will be signed by patient and their mainly caregiver.

Patient's QoL will be assessed using self-administered questionnaires Kidscreen 10 and VSP-A. In addition coping (KidCope), anxiety (STAI-C, STAI-Y), personality / attachment (IPPA), optimism (Y-LOT) measures and socio-demographic data will be collected. Self-administered questionnaires will be used for assessing caregivers' Qol (SF36), anxiety (STAI-Y), coping (BriefCope situational format), health care system satisfaction (Care quality scale) and burden (Zarit Caregiver Burden Inventory). Child's QoL evaluated by caregivers will be assessed using QUALIN, Kidscreen 10 parent and VSP-Ap. In addition, socio-demographic data, urban environment and economic environment will be collected. Clinical data will be collected by health professionals.

Results expected A sample of 136 children with ESRD is expected for identifying individual and populational factors which could influence chronic dialysed children QoL, in order to propose adjustments to optimize these patients quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Minors patients treated by dialysis or on standby of graft availability

Exclusion Criteria:

* Minors patients treated by dialysis for less than 4 weeks

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 136 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Numbers of patient with identicals factors influencing chronic dialysed children quality of life as assessed by Kidscreen 10 scales | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Michel TSIMARATOS, MD/PhD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No